CLINICAL TRIAL: NCT00293878
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Safety and Effects on Lipids of 12 Weeks of 2 Doses of FM-VP4 in Subjects With Primary Hypercholesterolemia
Brief Title: Study on the Safety and Effects on Lipids of FM-VP4 in Subjects With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forbes Medi-Tech (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL2005-001
Record Dates: First submitted 2006-01-17; First posted 2006-02-20 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2007-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — FM-VP4 compound

INTERVENTIONS:
Drug: Disodium Ascorbyl Phytostanol Phosphate (FM-VP4)

SUMMARY:
The purpose of this study is to evaluate the safety and effects on lipids of FM-VP4 administered for 12 weeks in subjects with mild to moderate primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate primary hypercholesterolemia
* Able to give informed consent and to comply with study procedures (including diet)

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Age <18 or >75 years
* Pregnant women or women of child-bearing potential

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-11

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C at 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline in TC, HDL-C, TG, HDL:LDL ratio and CRP at 12 weeks
Percent change from baseline in serum lipids at 2, 4 and 8 weeks
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jean Warner, MD, Study Director — Clinical Consultant
Locations (14):
- United States (14):
  - Coastal Clinical Research, Mobile, Alabama
  - Radiant Research, San Diego, California
  - Radiant Research, Daytona Beach, Florida
  - Radiant Research, Gainesville, Florida
  - Radiant Research, Boise, Idaho
  - Radiant Research, Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - PRA International Pharmacology Center, Lenexa, Kansas
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Radiant Research, Portland, Oregon
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Radiant Research, Austin, Texas
  - Research Across America, Dallas, Texas
  - Radiant Research, Dallas, Texas